CLINICAL TRIAL: NCT05932082
Title: The Impact of Myomectomy on IVF Outcomes: A Multicenter Randomized Controlled Trial
Brief Title: The Impact of Myomectomy on IVF Outcomes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MIO study
Record Dates: First submitted 2023-06-10; First posted 2023-07-06 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Myoma;Uterus; IVF; Surgery
MeSH Terms: conditions — Myofibroma | interventions — Uterine Myomectomy; Nuclear Receptor Subfamily 4, Group A, Member 2

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- myomectomy group (Experimental): The study group received IVF after myomectomy.
  Interventions: Procedure: myomectomy or not
- control group (Placebo Comparator): The control group was directed to IVF after the routine evaluation, probably including diagnostic laparoscopy.
  Interventions: Procedure: myomectomy or not

INTERVENTIONS:
Procedure: myomectomy or not — The study group receive myomectomy, while the control group don't receive myomectomy.

SUMMARY:
In 2% to 3% infertility women, myoma is the only factor relevant to their infertility. However, the effects of intramural myoma on fertility are controversial. For infertile women with intramural myoma (types IV, V, VI of FIGO system) of 4 to 6 cm diameter, it is not clear whether myomectomy could improve pregnancy outcomes, especially in women undergoing ART. Besides, rigorous clinical research is needed to explore the changes and relevant biomarkers of endometrial receptivity through multi-omics study in patients undergoing myomectomy and ART treatment.

Method Intervention and follow-up: (1) For the control group, evaluation protocols such as salpingography and/or laparoscopic tubal fluxation should be implemented to identify disorders such as hydrosalpinx. (2) Imaging evaluation: all pelvic MRI were performed. Other options such as transvaginal ultrasound are not excluded, but won't replace MRI. Enhanced MRI or DWI may be considered, but are not always required. (3) Surgical intervention: laparoscopic myomectomy is preferred, and abdominal myomectomy is also acceptable. (4) IVF treatment: the IVF regimen should include detailed records of the downregulation plan, number of cycles, frozen or fresh blastocysts.

Study endpoints

(1) Primary study endpoint: Live birth rate after IVF. (2) Secondary study endpoints: Clinical pregnancy rate after IVF; Cumulative pregnancy rate after IVF; Biochemical pregnancy rate after IVF; Sustained pregnancy rate after IVF (≥20 weeks); Miscarriage rate after IVF; Cycles of IVF; Pregnancy-related complications; Perinatal maternal and neonatal complications. (3) Exploratory endpoints: The correlation between imaging index and assisted reproductive outcomes, including endometrial thickness, uterine volume, type of endometrial echo, uterine contraction; endometrial vascular index (VI), flow index (FI), tubular flow index (VFI); uterine artery pulsation index (PI), uterine artery resistance index (RI), systolic/diastolic blood pressure of uterine artery (S/D).

The correlation between endometrial receptivity and assisted reproductive outcomes is analyzed based on transcriptomics, metabolomics, methylation and proteomics in samples from peripheral blood, endometrial biopsy, endometrial exfoliated cells, cervical exfoliated cells and myoma.

DETAILED DESCRIPTION:
Grouping and blinding method This is a national multicenter, randomized controlled study. Competitive enrollment is performed among all centers. The study group received IVF after myomectomy and the control group was directed to IVF after the routine evaluation, probably including diagnostic laparoscopy. In this study, 792 patients were randomly divided into 2 groups with 396 patients in each group according to centralized random system. A random sequence is generated with a random block size of a block size of 4.

Collection of clinical data and samples Data and samples are collected according to Case Report Form (CRF) form, including randomized information, epidemiologic and clinical information. Evaluation of infertility history and details, imaging results, ovarian reservation and surgical findings are of special interest and detailed recorded.

Samples of peripheral blood, cervical exfoliated cells, endometrial exfoliated cells, endometrial biopsy and myoma in study group are collected for multi-omics analysis. The process of sample harvest shouldn't interfere or deteriorate the surgical and IVF treatment.

IVF treatment: the IVF regimen should include detailed records of the downregulation plan, number of cycles, frozen or fresh blastocysts, ①Study group: IVF treatment is performed 6 months after myomectomy, and patients should be followed up for 1 year after the start of IVF. If the endometrium is exposed during myomectoy, IVF treatment is performed 12 months after myomectomy. It should be noted that the time for postoperative contraception should be recorded, and also the time interval between myomectomy and IVF.

②Control group: IVF treatment was performed immediately after relevant evaluation, and follow-up for 1 year after the start of IVF.

Genomic feature examination and bioinformatics analysis

1. Endometrial receptive array (ERA) is a molecular diagnostic test based on microarray technology, which divides endometrial biopsy into receptive, pre receptive, or proliferative types based on the expression of 238 selected genes. ER Map/ER Stage is based on the expression of 184 genes involved in maternal immune response related to endometrial proliferation and embryo implantation.
2. Methylation sequencing: Extract DNA related to peripheral blood, tissue, and cells, and accurately quantify DNA concentration using Qubit 2.0. The total amount of DNA detected should not be less than 1ug. Library construction: After passing the sample detection, 1 µ g of sample genomic DNA was mixed with unmethylated lambda DNA using the Biouptor system, and then fragmented to an average size of approximately 250bp. After fragmentation, the purified random fragmented DNA was then repaired, passivated and phosphorylated with a mixture of T4 DNA polymerase, Klenow fragment and T4 polynucleotide kinase. The blunt DNA fragment was then 3 'adenosylated with Klenow fragment (3' -5'exo -), and then linked to the linker connecting 5 '- methyl Cytosine instead of Cytosine using T4 DNA ligase. After completing each step, use magnetic beads to purify DNA. Then, use ZYMO EZ DNA methylation gold kit to convert unmethylated Cytosine to Uracil according to instructions. Finally, use JumpStart Taq DNA polymerase for PCR amplification, and then use magnetic beads to purify the PCR product to obtain the final library. Library quality inspection: After the construction of the library is completed, preliminary quantification is carried out using Qubit2.0, and the library is diluted to 1ng/ul. Then, the insert size of the library is tested using Agilent 2100. After the insert size meets expectations, the effective concentration of the library is accurately quantified using qPCR method (effective concentration of the library>2nM) to ensure library quality. Online sequencing: After passing the library detection, different libraries are pooled according to the effective concentration and target offline data volume requirements, and then sequenced on the Illumina Nova platform using the PE150 sequencing strategy. After that, quality control of original offline data, sequence comparison, calculation of methylation level, identification and statistics of differential methylation region (DMR) were carried out.

Urinary protein detection and bioinformatics analysis

1. Protein separation technology: two-dimensional gel electrophoresis (2DE), two-dimensional fluorescence differential electrophoresis (2D-DIGE), isoelectric focusing electrophoresis (IEF), liquid chromatography; Multidimensional chromatography (MDC) (including size exclusion chromatography, ion exchange chromatography, reverse phase high performance chromatography, hydrophobic interaction chromatography, etc.), and multidimensional liquid chromatography (MDLC).
2. Protein identification technology: primary mass spectrometry: according to different ion sources, it can be divided into matrix assisted laser desorption ionization time of flight mass spectrometry (MALDI-TOF-MS) and electric spray mass spectrometry (ESI MS); Secondary mass spectrometry: peptide mass fingerprint (PMF); New technology: Stable nuclide signature bio mass spectrometry (SIAMS).
3. Identification of protein peptide segments: amino and carboxyl end analysis, such as Edman; Mass spectrometry, including peptide fragment mass spectrometry and tandem mass spectrometry.
4. Protein interactions: Immunoprecipitation technology, Yeast two hybrid system, Protein chip technology.

Metabolomics and Bioinformatics Analysis

1. The endometrium tissue was immediately frozen in liquid nitrogen after being isolated, and then the tissue was stored at -80 ℃, ground and crushed, and extracted with cold organic Liquid-liquid extraction. Attention must be paid to avoiding metabolic changes before and during sampling. Perform metabolomics analysis on collected cells, tissues, blood, and urine.
2. Metabolite extraction: The most commonly used method in metabolite extraction is to precipitate protein with organic solvents, and extract the supernatant through high-speed centrifugation or ultrafast filtration to remove protein precipitation. Concentrate using freeze-drying or nitrogen blowing, and dissolve the residue in a complex solvent.
3. Sample detection: Take a certain amount of redissolved supernatant and use Thermo Vanquish UHPLC ultra-high performance liquid chromatography system and Thermo Q Active HF-X mass spectrometry platform for machine detection.
4. Data processing: After the mass spectrometry detection is completed, the offline data (. raw) file is imported into the search software for simple screening of retention time, mass charge ratio, and other parameters. Then, according to the retention time deviation, quality deviation and signal strength deviation, signal to noise ratio, minimum signal strength and other information of different samples, peak alignment and peak extraction are carried out. At the same time, the peak area is quantified, and then the target ions are integrated to predict the Molecular formula and compare with the database to obtain the identification and quantitative results of the data. Therefore, non targeted metabolomics databases and search software play a decisive role in the experimental results. However, LC-MS has very few public databases, and most of them are platform built databases. The commonly used databases include HMDB, METLIN, and some self built libraries.
5. Information analysis: Principal component analysis, differential metabolite analysis, etc.

ELIGIBILITY:
Inclusion Criteria:

1. Female aged between 20-40 years old.
2. Primary or secondary infertility consisting of following factors rather than uterine factors: male factors, ovulation disorders, fallopian tube factors, endometriosis, other non-uterine factors including infertility with unexplained reason.
3. Myoma: FIGO type 4-6 discovered by MRI with the maximum diameter surgically targeted between 4-6cm; Single myoma, or multiple myomas with non-surgically targeted intramural or subserous myoma(s) < 2cm in maximum diameter.
4. Justifying the IVF criteria and willing to undergo IVF.

Exclusion Criteria:

1. Not meeting all the inclusion criteria.
2. Complicated with infertility factors of uterine factors or diseases, including adenomyosis, endometrial adhesion, endometritis, submucous myoma. However, resectable endometrial polyps need not be excluded.
3. Complicated with malignancies or borderline tumors of the reproductive tract
4. Complicated with other malignancies not been treated or still being treated.
5. Complicated with active pelvic inflammatory disease.
6. Previously receiving cytotoxic therapy or abdominal-abdominal chemoradiotherapy.
7. Previous uterine body surgery, including but not limited to: myomectomy, resection for adenomyosis lesions, uterine artery embolization, uterine tumor coagulation (high energy focused ultrasound or electrocoagulation, hysteroscopically myomectomy. However, diagnostic hysteroscopy, diagnostic curettage and polypectomy need not be excluded.
8. No willing to undergo IVF.
9. Unable to be followed-up.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 792 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with live birth after IVF within one year | one year after IVF
  Live birth rate after IVF in infertility patients with intramural myoma (types IV, V, VI) with a diameter of 4-6cm receiving or not receiving myomectomy.

SECONDARY OUTCOMES:
Number of participants with of clinical pregnancy after IVF within one year | one year after IVF
  Clinical pregnancy rate after IVF in infertility patients with intramural myoma (types IV, V, VI) with a diameter of 4-6cm receiving or not receiving myomectomy.
Number of participants with cumulative pregnancy after IVF within one year | one year after IVF
  Cumulative pregnancy rate after IVF in infertility patients with intramural myoma (types IV, V, VI) with a diameter of 4-6cm receiving or not receiving myomectomy.
Number of participants with Biochemical pregnancy rate after IVF | one year after IVF
  Biochemical pregnancy rate after IVF in infertility patients with intramural myoma (types IV, V, VI) with a diameter of 4-6cm receiving or not receiving myomectomy.
Number of participants with sustained pregnancy rate after IVF (≥20 weeks) | at least 20 weeks after IVF
  Sustained pregnancy rate after IVF in infertility patients with intramural myoma (types IV, V, VI) with a diameter of 4-6cm receiving or not receiving myomectomy.
Number of participants with miscarriage after IVF | one year after IVF
  Miscarriage rate after IVF in infertility patients with intramural myoma (types IV, V, VI) with a diameter of 4-6cm receiving or not receiving myomectomy.
number of cycles of IVF | one year after IVF
  Cycles of IVF in infertility patients with intramural myoma (types IV, V, VI) with a diameter of 4-6cm receiving or not receiving myomectomy.
Number of participants with pregnancy-related complications | one year after IVF
  Pregnancy-related complications after IVF in infertility patients with intramural myoma (types IV, V, VI) with a diameter of 4-6cm receiving or not receiving myomectomy.
Number of participants with perinatal maternal and neonatal complications | one year after IVF
  Perinatal maternal and neonatal complications after IVF in infertility patients with intramural myoma (types IV, V, VI) with a diameter of 4-6cm receiving or not receiving myomectomy.